CLINICAL TRIAL: NCT04391920
Title: Registry of CytoSorb Therapy in COVID-19 ICU Patients (CTC REGISTRY): Registry of Patient-level Clinical Data on CytoSorb Hemoadsorption Provided Via Integration of the CytoSorb Device Into Extracorporeal Membrane Oxygenation (ECMO), Continuous Renal Replacement Therapy (CRRT), or Hemoperfusion Extracorporeal Circuits in COVID-19 ICU Patients
Brief Title: Registry of CytoSorb Therapy in COVID-19 ICU Patients
Acronym: CTC REGISTRY
Status: Completed | Type: Observational
Sponsor: CytoSorbents, Inc (Industry)
Collaborators: CytoSorbents Europe GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-001; FDA EUA (Other: FDA)
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- COVID-19 ICU Patients
  Interventions: Device: CytoSorb 300 mL device

INTERVENTIONS:
Device: CytoSorb 300 mL device — CytoSorb hemoadsorption provided via integration of the CytoSorb device into ECMO, CRRT, or hemoperfusion extracorporeal circuits.

SUMMARY:
The CTC Registry collects patient-level clinical data on CytoSorb hemoadsorption provided to COVID-19 ICU patients via integration of the CytoSorb device into ECMO, CRRT, or hemoperfusion extracorporeal circuits. The intent of the registry is to gain understanding on how CytoSorb hemoadsorption provides clinical benefit to COVID-19 ICU patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed COVID-19
2. Provision of CytoSorb therapy per Instructions for Use (IFU) of the CytoSorb device.

Exclusion Criteria:

1. CytoSorb therapy for diseases other than COVID-19
2. Survival unlikely within 24 hours (for prospectively enrolled patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 ICU patients receiving CytoSorb hemoadsorption via integration of the CytoSorb device into ECMO, CRRT, or hemoperfusion extracorporeal circuits.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
ICU mortality | From the date of start of CytoSorb use until the date of ICU discharge or date of death, whichever comes first, assessed up to 1 year

SECONDARY OUTCOMES:
Duration of ECMO after start of CytoSorb | From the date of start of CytoSorb use until the date of cessation of ECMO or date of death, which ever comes first, assessed up to 1 year
Duration of mechanical ventilatory support after start of CytoSorb | From the date of start of CytoSorb use until the date of cessation of mechanical ventilatory support or date of death, which ever comes first, assessed up to 1 year
Duration of pharmacologic hemodynamic support after start of CytoSorb | From the date of start of CytoSorb use until the date of cessation of pharmacologic hemodynamic support or date of death, which ever comes first, assessed up to 1 year
Change in serum concentrations of inflammatory biomarkers after start of CytoSorb | From the day before start of CytoSorb use until the day after cessation of CytoSorb use
Change in Pa02/Fi02 ratio after start of CytoSorb | From the day before start of CytoSorb use until the day after cessation of CytoSorb use

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nelson, MD, Study Director — CytoSorbents Corporation
Locations (7):
- United States (7):
  - Medical Center of Aurora, Aurora, Colorado
  - University of Chicago Medicine, Chicago, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Baptist Memorial Hospital, Southaven, Mississippi
  - New York University Medical Center, New York, New York
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hayanga JWA, Song T, Durham L, Garrison L, Smith D, Molnar Z, Scheier J, Deliargyris EN, Moazami N. Extracorporeal hemoadsorption in critically ill COVID-19 patients on VV ECMO: the CytoSorb therapy in COVID-19 (CTC) registry. Crit Care. 2023 Jun 19;27(1):243. doi: 10.1186/s13054-023-04517-3. PMID 37337243
- [Derived] Song T, Hayanga J, Durham L, Garrison L, McCarthy P, Barksdale A, Smith D, Bartlett R, Jaros M, Nelson P, Molnar Z, Deliargyris E, Moazami N. CytoSorb Therapy in COVID-19 (CTC) Patients Requiring Extracorporeal Membrane Oxygenation: A Multicenter, Retrospective Registry. Front Med (Lausanne). 2021 Dec 20;8:773461. doi: 10.3389/fmed.2021.773461. eCollection 2021. PMID 34988092